CLINICAL TRIAL: NCT04163588
Title: Early Sequential Nephron Blockade Versus Standard Diuretic Treatment in Acute Heart Failure
Brief Title: Sequential Nephron Blockade in Acute Heart Failure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Policlinico Casilino ASL RMB (Other)
Collaborators: Umberto I Hospital, Nocera Inferiore (Other); IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Leonardo Calò, MD, Professor, Policlinico Casilino ASL RMB
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNB01
Record Dates: First submitted 2019-10-26; First posted 2019-11-15 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Acute Heart Failure
Keywords: acute heart failure; decongestion; diuretics; outcomes
MeSH Terms: interventions — Metolazone; Sodium Potassium Chloride Symporter Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard therapy (Active Comparator): intravenous loop diuretics as recommended by current guidelines plus placebo
  Interventions: Drug: Loop Diuretics
- SNB (Experimental): loop diuretics plus oral metolazone at a dose of 5/10 mg once daily
  Interventions: Drug: Metolazone; Drug: Loop Diuretics

INTERVENTIONS:
Drug: Metolazone — Study participants receive loop diuretics plus oral metolazone at a dose of 5/10 mg once daily
  Arms: SNB
Drug: Loop Diuretics — Study participants receive a standard diuretic strategy (intravenous loop diuretics as recommended by current guidelines plus placebo)

SUMMARY:
Background - Volume overload is an important clinical target in acute heart failure management (AHF), typically addressed using loop diuretics. An important and challenging subset of heart failure patients exhibit fluid overload despite significant doses of loop diuretics. One approach to overcome loop diuretic resistance is the addition of a thiazide-type diuretic to produce diuretic synergy via "sequential nephron blockade". Although potentially able to induce diuresis in patients otherwise resistant to high doses of loop diuretics, this strategy has not been subjected to large-scale clinical trials to establish safety and clinical efficacy.

Methods - Our trial is a multicentric, double blind, randomized clinical study, aiming to recruit 310 patients with AHF and clinically evident volume overload. Study participants are randomized to receive a standard diuretic therapy (intravenous loop diuretics as recommended by current guidelines plus placebo) or SNB therapy (loop diuretics plus oral metolazone at the dose of 5/10 mg once daily) on top of standard medical therapy. Mineralocorticoid antagonists will be used in association with the two regimens according to blood potassium level and kidney function at the discretion of the treating physician. The primary endpoint is defined as the change in the serum creatinine level and the change in weight, considered both as a bivariate response and with their single components, between the time of randomization and 72 hours after randomization. Secondary endpoints include global well-being and dyspnoea assessed by a visual-analogue scale, changes in body weight and net fluid loss, proportion of patients free from congestion, treatment failure, changes in biomarker levels and the composite of death, rehospitalization, or an emergency room visit within 60 days, as well as the composite of total number of days hospitalized or death during the 60 days after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent must be obtained before any study assessment is performed
* Male or female patients 18 years of age or older
* An elective or emergency hospital admission with clinical diagnosis of decompensated HF with at least one clinical sign of volume overload (e.g. oedema (score 2 or more), ascites confirmed by echography or pleural effusion confirmed by chest X-ray or echography) Plasma NT-proBNP levels >1000 ng/mL or BNP levels >250 ng/mL at the time of screening.

Assessed LVEF by any imaging technique; i.e. echocardiography, catheterization, nuclear scan or magnetic resonance imaging within 12 months of inclusion

Exclusion Criteria:

* Concurrent diagnosis of an acute coronary syndrome defined as typical chest pain in addition to a troponin rise above the 99th percentile and/or electrocardiographic changes suggestive of cardiac ischemia
* History of congenital heart disease requiring surgical correction
* History of a cardiac transplantation and/or ventricular assist device
* Systolic blood pressure <90 mmHg or mean arterial pressure <65 mmHg at the moment of admission
* Estimated glomerular filtration rate <20 mL/min/1.73m² at screening
* Use of renal replacement therapy or ultrafiltration at any time before study inclusion
* Treatment with metolazone during the index hospitalization and prior to randomization
* Exposure to nephrotoxic agents (i.e. contrast dye) anticipated within the next 3 days
* Use of any non-protocol defined diuretic agent with the exception of mineralocorticoid receptor antagonists.
* Current use of sodium-glucose transporter-2 inhibitors
* Subjects who are pregnant or breastfeeding

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
change in the serum creatinine level and the change in weight, considered both as a bivariate response and with their single components | 72 hours
  The bivariate response will be displayed on a two-dimensional grid with individual data points for each patient representing paired changes in both creatinine (inmg/dL) and weight (in kilograms) 76 hours after randomization. A confidence region for the average difference between treatment arms in this bivariate response can be described as an ellipse, and the 2 treatment arms will be compared statistically with the use of the Hotelling T- square, which is a multivariate analog of the 2-sample t test used with a single continuous variable (Ann Math Stat. 1931; 2:360-78). Evaluating these 2 important responses to treatment as a bivariate end point reflects clinically important responses to therapy and avoids the requirement of making adjustments in sample size to prevent a type 1 error that would be necessary if the end points were considered separately (Eur J Heart Fail. 2003; 5:717-23).

SECONDARY OUTCOMES:
global well-being assessment by a visual-analogue scale | 72 hours
  Global well-being is assessed with the use of a visual-analogue scale that ranged from 0 to 100, with higher scores indicating greater well-being (Chest 1999;116:1208-17)
body weight assessment | 72 hours
  total changes in body weight in kilograms
congestion | 72 hours
  proportion of patients who were free from congestion (defined as jugular venous pressure of <8 cm, with no orthopnoea and with trace peripheral oedema or no oedema)
treatment failure | 7 days
  death, worsening/persistent HF, need for dialysis, crossover from standard pharmacologic care to sequential nephron blockade or the occurrence of a serious adverse event during the first 7 days from admission
Biomarkers | 72 hours, 7 days or discharge
  changes in NT-proBNP levels (in pg/mL) at 72 hours, day 7 or discharge
clinical end-point | 60 days
  composite of death, rehospitalization, or an emergency room visit within 60 days
hospitalization-death | 60 days
  composite of total number of days hospitalized or dead during the 60 days after randomization
Total net fluid loss | 76 hours
  total urinary output (in milliliters) from randomization to 76 hours
dyspnea assessment by a visual-analogue scale | 76 hours
  Dyspnea is assessed with the use of a visual-analogue scale that ranged from 0 to 100, with higher scores indicating less dyspnea (Chest 1999;116:1208-17)

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Cice, MD, Principal Investigator — Policlinico Casilino
Locations (1):
- Policlinico Casilino, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Undecided